CLINICAL TRIAL: NCT01098916
Title: The RAD-HOME Project: a Randomized Pilot Study of a Domiciliary Teleradiology Program for Frail Elderly Patients
Brief Title: The RAD-HOME Project: a Pilot Study of Domiciliary Teleradiology
Acronym: RHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Collaborators: FondazioneCRT (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0078572
Record Dates: First submitted 2010-03-10; First posted 2010-04-05 (Estimated); Last update posted 2010-04-05 (Estimated); Status verified 2008-05

CONDITIONS: Acute Congestive Heart Failure; Exacerbation of COPD; Pneumonia; Fractures; Osteomyelitis
Keywords: hospital at home; radiology at home; frail elderly
MeSH Terms: conditions — Pneumonia; Fractures, Bone; Osteomyelitis | interventions — X-Rays; Hospitals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- X-rays at home (Experimental): Home hospitalized elderly patients undergo X-rays at home
  Interventions: Radiation: Home X-rays
- Hospital X-rays (Active Comparator): Home hospitalized elderly patients undergo X-rays examinations in hospital
  Interventions: Radiation: X-rays in hospital

INTERVENTIONS:
Radiation: Home X-rays — X-rays examinations performed at home
  Arms: X-rays at home
Radiation: X-rays in hospital
  Arms: Hospital X-rays

SUMMARY:
Aim of the study is to assess feasibility and safety of a public territorial radiology service for home hospitalized frail elderly patients whose health conditions discourage the transportation to hospital.

ELIGIBILITY:
Inclusion Criteria:

* immobilization or chairbound,
* need for chest, pelvis/hips, joints, upper and lower limbs, hands and feet X-rays,
* absence of definite delirium at enrollment according to the Confusion Assessment Method, and
* intermediate or high risk of delirium according to the criteria of Inouye.

Exclusion Criteria:

* need of urgent examination (within 24 hours),
* need of X-ray examinations not suitable at home.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Comparison of episodes of delirium related to the radiological procedure at home and in hospital, using the Confusion Assessment Method (CAM) | 24 hours after the radiological procedure
  Frail patients, especially old ones,often develop delirium or confusion when moved from their usual environment. In home-hospitalized patients with the same risk of developing delirium, according to the Inouye's criteria, we evaluated the onset of a confusional status after X-rays performed at home or in hospital

SECONDARY OUTCOMES:
Evaluation of direct and indirect costs of the radiological procedures performed at home or in hospital | 1 year
  Evaluation of costs includes: costs for transportation, ambulance, equipment (eg, processing costs), materials (eg, CD), technical staff (eg, radiographers, radiologists); for the control group: costs for working time employed by family members and health staff to bring patients to hospital for X.ray examination
Satisfaction of patients and/or families | within 1 month after the procedure
  Customer satisfaction is evaluated using an ad hoc questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Cammarota, MD, Principal Investigator — Fifth Radiology Department, San Giovanni Battista Hospital of Torino
Locations (1):
- San Giovanni Battista Hospital, Torino, Italy

REFERENCES:
- [Derived] Ricauda NA, Tibaldi V, Bertone P, Quagliotti E, Tizzani A, Zanocchi M, Isaia GC, Grosso M, Cammarota T, Davini O. The RAD-HOME project: a pilot study of home delivery of radiology services. Arch Intern Med. 2011 Oct 10;171(18):1678-80. doi: 10.1001/archinternmed.2011.336. Epub 2011 Aug 8. No abstract available. PMID 21824941